CLINICAL TRIAL: NCT02547701
Title: Multicentre, Open Label Study to Assess the Tolerability of P-3058 Nail Solution in Paediatric Patients Affected by Mild-to-moderate Onychomycosis
Brief Title: Clinical Trial on Onychomycosis With P-3058 Nail Solution in Pediatric Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polichem S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM Ped-004; 2013-005595-17 (EudraCT Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-11 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P-3058 (Experimental)
  Interventions: Drug: P-3058

INTERVENTIONS:
Drug: P-3058

SUMMARY:
Pediatric patients affected by mild-to-moderate distal subungual onychomycosis (DSO) or affected by white superficial onychomycosis (WSO), due to dermatophytes, will be treated topically with P-3058 nail solution according to the appropriate treatment schedule.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 to 17 years
* Males and females
* Clinical diagnosis of mild-to-moderate distal sub-ungual onychomycosis without spikes/dermatophytoma and without lunula involvement or white superficial onychomycosis.
* Positive mycroscopy examination from the target nail at screening.
* Positive culture for dermatophyte from the target nail at screening.

Exclusion Criteria:

* Patients with onychomycosis caused by yeasts or non-dermatophytes mould.
* Patients with nail psoriasis.
* Patients with nail changes due to eczema, lichen planus or alopecia areata.
* Patients with one-hand two-foot syndrome.
* Patients with immunodeficiency disorder or use of immune suppressive therapy 3 months prior to screening visit or need for it.
* Use of systemic antifungal drugs in the 6 months prior to screening visit.
* Use of topical nail antifungal drugs in the four weeks prior to screening visit.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Local tolerability | from week 4 up to maximum week 48 of treatment
  Local tolerability at all treated nails by means of the Severity Score for Skin Irritation

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Caserini, MD, Study Director — Polichem SA
Locations (5):
- Polichem Investigative site, One Investigational Site, Belgium
- Polichem Investigative Site, One Investigational Site, Germany
- Polichem Investigative site, One Investigational Site, Italy
- Polichem Investigative Site, One Investigational Site, Latvia
- Polichem Investigative Site, One Investigational Site, Spain